CLINICAL TRIAL: NCT05879367
Title: An Open-label, Phase 1b Study to Evaluate the Safety and Tolerability of Eflornithine Plus Temozolomide in Patients With Newly Diagnosed Glioblastoma or Astrocytoma
Brief Title: Evaluation of Eflornithine Plus Temozolomide in Patients With Newly Diagnosed Glioblastoma or Astrocytoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Orbus Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OT-21-101
Record Dates: First submitted 2023-05-03; First posted 2023-05-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma, IDH-wildtype; Glioblastoma; Glioblastoma Multiforme; Glioblastoma IDH (Isocitrate Dehydrogenase) Wildtype; GBM; Astrocytoma; Astrocytoma, IDH-Mutant
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Eflornithine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Eflornithine Dose Level 1 + Temozolomide (Experimental)
  Interventions: Drug: Eflornithine (Dose Level 1); Drug: Temozolomide
- Eflornithine Dose Level 2 + Temozolomide (Experimental)
  Interventions: Drug: Eflornithine (Dose Level 2); Drug: Temozolomide
- Eflornithine Dose Level -1 + Temozolomide (Experimental)
  Interventions: Drug: Eflornithine (Dose Level -1); Drug: Temozolomide

INTERVENTIONS:
Drug: Eflornithine (Dose Level 1) — Eflornithine 2.3 g/m2 administered orally every 8 hours on a 2 weeks on, 2 weeks off schedule
  Other Names: DFMO
  Arms: Eflornithine Dose Level 1 + Temozolomide
Drug: Eflornithine (Dose Level 2) — Eflornithine 2.8 g/m2 administered orally every 8 hours on a 2 weeks on, 2 weeks off schedule
  Other Names: DFMO
  Arms: Eflornithine Dose Level 2 + Temozolomide
Drug: Eflornithine (Dose Level -1) — Eflornithine 1.75 g/m2 administered orally every 8 hours on a 2 weeks on, 2 weeks off schedule
  Other Names: DFMO
  Arms: Eflornithine Dose Level -1 + Temozolomide
Drug: Temozolomide — Temozolomide 150 mg/m2 (with option to escalate per USPI maintenance phase instructions) administered orally once daily on a 5 days on, 23 days off schedule
  Other Names: Temodar; TMZ

SUMMARY:
The purpose of this study is to establish the recommended phase 2 dose of eflornithine in combination with temozolomide in patients whose glioblastoma or astrocytoma is newly diagnosed, and to evaluate safety and tolerability of this combination at that dose.

DETAILED DESCRIPTION:
This open label dose escalation and expansion study will be conducted using a standard dose-escalation design with escalating doses of eflornithine plus temozolomide at the approved dose level, followed by an expansion cohort that will further evaluate safety and preliminary efficacy of the combination at the recommended phase 2 dose.

Duration of participation will be up to approximately 104 weeks in total per patient.

Screening Period - A maximum screening duration of 4 weeks.

Treatment Period - Up to approximately 104 weeks.

Follow-Up Visit - 4 weeks from last treatment.

Long-term Survival Follow-Up - up to 2 years from last treatment.

A total of up to 66 patients will be enrolled in a non-randomized fashion (patients may be added to any of the dose levels below the RP2D to a maximum of approximately 20 per dose level with the intent of further characterizing safety and pharmacokinetics).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of World Health Organization (WHO) G4 classified GBM, IDH-wildtype (patients with GBM) or G3 astrocytoma (IDH1 or 2 mutant; CDKN2A/B intact) per WHO 2021 tumor classification.
* Completed external beam radiation therapy per standard of care.
* Patients with GBM: Must have received at least 80% of planned daily doses of TMZ during chemoradiation. Patients with astrocytoma: Must have tolerated adjuvant TMZ treatment through at least 2 and not more than 4 cycles.
* Adequate hematologic, renal, hepatic, and other organ function as indicated by hematology and serum chemistry testing.
* Willing to abstain from intercourse or use acceptable contraceptive methods.
* If taking corticosteroids, must be on a stable or decreasing dose.

Exclusion Criteria:

* Recent history of recurrent or metastatic cancer that could confound response assessments
* Prior systemic chemotherapy other than temozolomide during external beam radiation therapy (for patients with GBM) or adjuvant temozolomide through up to 4 pre-study cycles (for patients with astrocytoma).
* Prior Optune treatment.
* Active infection or serious intercurrent medical illness.
* Poorly controlled seizures.
* Significant cardiac disease within 6 months of enrollment.
* Poorly controlled diabetes.
* Use of another investigational agent within 30 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Dose Limiting Toxicities | 8 weeks
  Protocol Defined Dose Limiting Toxicities
Incidence of TEAEs All Grades | From enrollment to the follow-up visit 4 weeks after end of treatment
  All Grades
Incidence of TEAEs Grade 3+ | From enrollment to the follow-up visit 4 weeks after end of treatment
  Grade 3+
Incidence of TEAEs Serious | From enrollment to the follow-up visit 4 weeks after end of treatment
  Serious
Incidence of TEAEs Leading to Discontinuation | From enrollment to the end of treatment
  Leading to Discontinuation
Vital Signs (Heart and Respiratory Rate) | From enrollment to the follow-up visit 4 weeks after end of treatment
  Change from Baseline in Heart Rate and Respiratory Rate
Vital Signs (Blood Pressure) | From enrollment to the follow-up visit 4 weeks after end of treatment
  Change from Baseline in Systolic Blood Pressure and Diastolic Blood Pressure
Incidence of Treatment-Emergent Abnormalities in Clinical Laboratory Tests | From enrollment to the follow-up visit 4 weeks after end of treatment
  Lab abnormalities by CTCAE v5.0 Grade

SECONDARY OUTCOMES:
Overall Survival | From enrollment to up to 2 years after last dose
  Until death or initiation of new anticancer therapy
Progression Free Survival | From enrollment to the follow-up visit 4 weeks after end of treatment
  Per RANO Criteria as assessed by MRI
Overall Response Rate | From enrollment to the follow-up visit 4 weeks after end of treatment
  Per RANO Criteria as assessed by MRI
Pharmacokinetics Cmax | Baseline to Steady State (2 weeks)
  observed maximum concentration
Pharmacokinetics Cmin | Baseline to Steady State (2 weeks)
  observed minimum concentration
Pharmacokinetics Tmax | Baseline to Steady State (2 weeks)
  time of observed maximum concentration
Pharmacokinetics AUCt | Baseline to Steady State (2 weeks)
  area under the concentration-time curve
Pharmacokinetics lambdaz | Baseline to Steady State (2 weeks)
  elimination rate constant
Pharmacokinetics t 1/2 | Baseline to Steady State (2 weeks)
  elimination half life
QTcF-Concentration Relationship | Baseline to Steady State (2 weeks)
  Assessment of change in QTcF relative to plasma concentration of eflornithine
Assessment of QTcF | Baseline to Steady State (2 weeks)
  Change from baseline in QTcF

CONTACTS AND LOCATIONS:
Overall Officials: Howard Colman, MD, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Henry Ford Hospital, Detroit, Michigan
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Duke University, Durham, North Carolina
  - The Cleveland Clinic, Cleveland, Ohio
  - Brown University Health/Rhode Island Hospital, Providence, Rhode Island
  - UT MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No